CLINICAL TRIAL: NCT06278662
Title: Cohort Multiple Randomized Controlled Trial in Pediatric Asthma: Infrastructure to Assess the Long- and Short-term Effects of (eHealth) Interventions.
Brief Title: Cohort Multiple Randomized Controlled Trial in Pediatric Asthma
Acronym: CIRCUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mattienne van der Kamp (Other)
Responsible Party: Sponsor-Investigator, Mattienne van der Kamp, dr., Medisch Spectrum Twente
Organization: Medisch Spectrum Twente (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CIRCUS cmRCT
Record Dates: First submitted 2024-02-12; First posted 2024-02-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Pediatric Asthma
Keywords: asthma; child; cohort studies; telemedicine
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: The CIRCUS study has a cmRCT design to determine the effects of (eHealth) interventions in asthmatic children. Children are included in the prospective dynamic cohort during outpatient visits. Children and/or their parents are asked to sign consent for three parts of the cmRCT, of which at least consent for part 1 is needed to be eligible for participation:
  1. Participating in the prospective dynamic cohort and data collection.
  2. Willingness to participate in interventions.
  3. Willingness to fill out additional questionnaires and/or do additional measurements if a child is randomly selected for the control group of an intervention, which uses additional outcomes.
Masking Description: The masking is dependent of the future interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): The cohort multiple Randomised Controlled Trial (also known as TwiCs 'trials within cohorts') is a prospective study design in which (eHealth) intervention arms will be established over time. The interventions will be evaluated on the primary outcome measures of the cohort.
  Interventions: Other: video directly observed therapy (vDOT)
- Cohort control group (No Intervention)

INTERVENTIONS:
Other: video directly observed therapy (vDOT) — The first intervention of within the CIRCUS study is video directly observed therapy (vDOT). The intervention consists of taking recording of daily inhalation use and receiving four feedback sessions of an asthma nurse based on these home recordings.
  Arms: Intervention arm

SUMMARY:
The overarching goal of this study is to optimize pediatric asthma care and to continuously evaluate variations/innovations of the care (including transformation to remote eHealth care).

Primary Objectives within cmRCT cohort:

* Provide a framework for multiple randomized (eHealth) interventions for asthmatic children
* Generate short- and long-term data on Quality of life (QoL), asthma outcomes (asthma control, lung function), quality of care, self-management capacity, healthcare use, and therapy compliance in a representative secondary care pediatric asthma cohort.

Secondary Objectives within cmRCT cohort:

* Evaluate current pediatric asthma care at the Pediatric department of Medisch Spectrum Twente, in order to explore possible improvements for the pediatric asthma care.
* Compare the short and long-term asthma outcomes between the eHealth care path and the outpatient care path.
* Compose patient risk profiles that include both personal, clinical and exposome markers and clinical asthma endpoints (for example clinical admission/exacerbations).

DETAILED DESCRIPTION:
Rationale: Testing of eHealth interventions seems crucial since eHealth provides possibilities to obtain a real-time and objective view of asthma symptoms. Traditional randomized controlled trials(RCTs) face challenges in evaluating the effect of multiple eHealth components separately and in the long process of translating intervention ideas into funded research protocols, which may risk the eHealth intervention becoming outdated.

Objective: This study aims to provide a framework to assess the effect of (eHealth) interventions and generate short- and long-term data on clinical and patient-reported outcomes of asthmatic children using a cohort multiple Randomized Controlled Trial (cmRCT) design.

Study design: The CIRCUS study is a cmRCT designed to test multiple eHealth interventions in eligible asthmatic children (4-18 years old, treated in MST) within a cohort. Observational clinical data is collected of these children and both the children and their parents regularly complete questionnaires. In addition, a random selection of eligible children is approached for participation in interventions while the non-selected children remain in the control group.

Study population: Included children are 4-18 years old, diagnosed with asthma following the Global Initiative for Asthma (GINA) criteria and treated in Medisch Spectrum Twente at Enschede.

Main study parameters/endpoints: Primary outcome measures are Quality of life(QoL), asthma outcomes(asthma control, lung function), quality of care, self-management capacity, healthcare use, and therapy compliance.

Nature and extent of the burden and risks associated with participation, benefit, and group relatedness: Children and parents fill out questionnaires on a monthly and half-yearly basis. The questionnaires include: (C)-ACT, PAQLQ, CSQ-4, and PAM-13. In consultation with the patient panel we chose the shortest validated questionnaires to reduce the study burden. Other data (for example healthcare use) is collected by the researchers. No relevant risks were found in the risk analysis. We chose to use this group of children in this study as asthma management in children differs from that in adults.

ELIGIBILITY:
Inclusion Criteria:

* Is 4 to 18 years old
* Is patient at the children's department at Medisch Spectrum Twente at moment of inclusion
* Is diagnosed with asthma by a pediatrician following the Global Initiative for Asthma(GINA) guidelines 2022 [8]:

  *Medical history fitting asthma diagnosis:
* Based on (typical) symptoms: (nighttime) wheezing, dyspnea, coughing (triggered by either viral infections, exercise, allergens or weather changes)
* (Possibly) supplemented with a family history/atopy

AND

*Spirometry variable expiratory airflow limitation by at least one of these criteria:

* FEV1/FVC reduced compared to lower limit of normal(Z-score ≤ -1.64)
* Positive bronchodilator responsiveness(increase FEV1>12%)
* Positive Exercise Challenge Test (ECT)(decrease FEV1≥ 13%)
* Excessive variation in lung function (LF) between tests from different dates (variation FEV1>12% pred)

Exclusion Criteria:

* The child and/or parent(s) has/have insufficient command of the Dutch language resulting in the insufficient ability to understand and/or answer questions

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2034-04-01 (Estimated); Study Completion 2034-04-01 (Estimated)

PRIMARY OUTCOMES:
Asthma control | monthly (until the patient turns 18 years old, has no astma diagnosis anymore or is no longer under treatment of the MST hospital, whichever came first, assessed up to 168months)
  C-ACT/ACT: (Childhood) Asthma Control Test
Pediatric Asthma Quality of Life | once per 6 months (until the patient turns 18 years old, has no astma diagnosis anymore or is no longer under treatment of the MST hospital, whichever came first, assessed up to 168months)
  Pediatric Asthma Quality of Life Questionnaire (PAQLQ)
Quality of care | once per 6 months (until the patient turns 18 years old, has no astma diagnosis anymore or is no longer under treatment of the MST hospital, whichever came first, assessed up to 168months)
  CSQ-4: Client Satisfaction Questionnaire.
Self-management capacity | once per 6 months (until the patient turns 18 years old, has no astma diagnosis anymore or is no longer under treatment of the MST hospital, whichever came first, assessed up to 168months)
  PAM-13: patient activation measurement
Healthcare use | continuous (until the patient turns 18 years old, has no astma diagnosis anymore or is no longer under treatment of the MST hospital, whichever came first, assessed up to 168months)
  hospital admissions, outpatient visits, telephonic consultations, diagnostics,
Wheather data | daily (until the patient turns 18 years old, has no astma diagnosis anymore or is no longer under treatment of the MST hospital, whichever came first, assessed up to 168months)
  Wheather data (hourly): Temperature, humidity, rainfall
Air quality | daily (until the patient turns 18 years old, has no astma diagnosis anymore or is no longer under treatment of the MST hospital, whichever came first, assessed up to 168months)
  Hourly data on: Nitrogen dioxide(NO2), Nitric oxide(NO), Ozone(O3), Particulate matter(PM10), Particulate matter(PM2.5), Ultra Fine Particles(UFP) Carbon monoxide(CO2), Sulpher dioxide(SO2) Pollencount (daily): birch, grasses etc.
Pollen | daily (until the patient turns 18 years old, has no astma diagnosis anymore or is no longer under treatment of the MST hospital, whichever came first, assessed up to 168months)
  Pollencount (daily): Treepolls (Birch, Hazel, Alder, etc...) & bushes/grasspolls (grass, worm-wood, ambrosia, goose grass etc....)
Medication delivery | continous (until the patient turns 18 years old, has no astma diagnosis anymore or is no longer under treatment of the MST hospital, whichever came first, assessed up to 168months)
  LSP list via pharmacy of Medisch Spectrum Twente
  * Name medicine
  * Date of issue
  * Dose
  * Expected period of use
  * Quantity provided

CONTACTS AND LOCATIONS:
Locations (1):
- Medisch Spectrum Twente, Enschede, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruuls T, Sprengers R, Hengeveld V, Thio B, Tabak M, Zagers D, van der Palen J, van der Kamp M. Cohort multiple randomized controlled trial in pediatric asthma to assess the long- and short-term effects of eHealth interventions: protocol of the CIRCUS study. Ther Adv Respir Dis. 2025 Jan-Dec;19:17534666251323192. doi: 10.1177/17534666251323192. Epub 2025 Mar 12. PMID 40071339